CLINICAL TRIAL: NCT05595590
Title: Phase II Trial of Pulsed Radiotherapy Combined With Tislelizumab in Patients With Locoregionally Recurrent Head and Neck Squamous Cell Carcinoma
Brief Title: Radiotherapy With Tislelizumab in Patients With Recurrent Head & Neck Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20220816
Record Dates: First submitted 2022-10-19; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab + Pulse radiation (Experimental): Participants receive pulsed radiationtherapy concurrent with 3 cycles of Tislelizumab followed by an additional 32 cycles of Tislelizumab alone as maintenance therapy.
  Interventions: Drug: Tislelizumab; Radiation: Pulse radiation

INTERVENTIONS:
Drug: Tislelizumab — Administered as an intravenous (IV) infusion 200mg every 3 weeks (Q3W)
Radiation: Pulse radiation — 66-70Gy/33-35Fx, 2Gy/Fx.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of pulsed radiotherapy given concomitantly with Tislelizumab and as maintenance therapy in participants with locoregionally recurrent head and neck squamous cell carcinoma ( HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed squamous cell head and neck cancer, A karnofsky performance status≥70.
* Previous radical therapy (surgery ± chemoradiotherapy or radical chemoradiotherapy) and the records of radiation fields and dosage of previous treatment can be obtained.
* Inoperable or completely resectable under MDT consultation.
* Has evaluable tumor burden (measurable and/or non-measurable tumor lesions) assessed by computed tomography scan or magnetic resonance imaging, based on RECIST version 1.1
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study therapy
* Female and male participants of reproductive potential must agree to use adequate contraception throughout the study period and for up to 180 days after the last dose of study therapy

Exclusion Criteria:

* Pregnant or breastfeeding, or planning to become pregnant during the study period
* The patient had another malignant tumor expcet HNSCC
* Have an active autoimmune disease or immunodeficiency, including but not limited to myasthenia gravis, interstitial pneumonia, enteritis, autoimmune hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, test positive for HIV or have a history of any of these diseases, or have a history of organ transplantation;
* They had received reradiotherapy within 1 month prior to entering the study
* Receiving systemic immunosuppressive drugs within 2 weeks prior to commencing study treatment, or anticipating needing systemic immunosuppressive drugs during study treatment;
* having received systemic immune-stimulating agents (including but not limited to interferon or interleukin-2 [IL-2]) within 4 weeks prior to study treatment initiation or remaining within 5 half-lives (whichever is longer);
* A history of other malignancies within the past 5 years, except cured cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, and ductal carcinoma in situ;
* Severe cardiovascular disease (e.g., New York College of Cardiology heart disease class Ⅱ or greater, myocardial infarction, or cerebrovascular accident), unstable arrhythmia, or unstable angina within 3 months before commences study treatment;
* The subject has an active infection or infectious disease, or develops a fever of unknown origin (body temperature >38.5 ° C) during screening and before the first dose;
* had received therapeutic oral or intravenous antibiotics within 2 weeks prior to starting the study; Patients receiving prophylactic antibiotic therapy, such as prevention of urinary tract infection or chronic obstructive pulmonary disease, were enrolled.
* Untreated active hepatitis (hepatitis B: HBsAg positive with abnormal liver function and HBV-DNA≥104ml; Hepatitis C: HCV-RNA≥103/ml or antiviral therapy required during the study);
* Immunotherapy such as PD-1/L1 antibody or CTLA-4 antibody within 4 weeks before enrollment.
* Chemotherapy or targeted therapy within 4 weeks prior to enrollment;
* Subjects have participated in or completed other clinical trials within 4 weeks prior to enrollment;
* Subjects may need to receive other antitumor treatments during the study;
* Subjects may need to have been vaccinated during the study or within 4 weeks prior to enrollment.
* A patient who, in the investigator's judgment, has other comorbidities that seriously jeopardize the patient's safety or interfere with the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2024-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) using iRECIST 1.1 criteria | From time of first dose of study treatment until disease progression or death (up to 2 years)
  ORR is defined as the proportion of patients who achieved a best response of complete response (CR) or partial response (PR) using iRECIST 1.1 criteria, and will be evaluated for both the lesion(s) treated with RT, referred to as "Target lesion (RT+ Tisle), as well as the lesion(s) not treated with RT (if applicable), referred to as "Target lesion (Tisle only)", per the prescribed treatment.
Adverse Events (AEs) | From time of first dose of study treatment until the end of follow-up (up to 2 years)
  Number of participants experiencing any sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study therapy.

SECONDARY OUTCOMES:
Duration of Response (DOR) | From time of first dose of study treatment until disease progression or death (up to 2 years)
  The time between the date of first confirmed response to the date of the first documented tumor progression, or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) | From time of first dose of study treatment until disease progression or death (up to 2 years)
  PFS is the average length of time after the start of treatment in which a person is alive, and their cancer does not grow or spread. PFS is defined as the time from day 1 of treatment until the criteria for disease progression is met as defined by RECIST1.1 or death as a result of any cause.
Change From Baseline Quality of Life (GHS/QoL) | From time of first dose of study treatment until disease progression or death (up to 2 years)
  Change from baseline in QoL using the European Organization for Research and Treatment of Cancer Head and Neck Questionnaire (EORTC QLQ-H&N35)

CONTACTS AND LOCATIONS:
Overall Officials: Ximei Zhang, Dr., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (2):
- China (2):
  - Sichuan Cancer Hosiptal, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No